CLINICAL TRIAL: NCT01375803
Title: Novel Fiber Effects on Glucose Metabolism and Insulin Sensitivity for Individuals at High Risk for Diabetes
Brief Title: Effects of Novel Fiber on Glucose Metabolism and Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cargill (Industry)
Responsible Party: Anne Franck, PhD, Cargill Incorporated
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CFIS-09-001
Record Dates: First submitted 2011-06-16; First posted 2011-06-17 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2011-06

CONDITIONS: Insulin Resistance
Keywords: dietary fiber; fiber; insulin sensitivity; insulin resistance; glucose metabolism
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): 3g/day
  Interventions: Dietary Supplement: Novel dietary fiber
- 2 (Experimental): 6g/day
  Interventions: Dietary Supplement: Novel dietary fiber
- Placebo beverage (Placebo Comparator): 0g/day
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Novel dietary fiber — oral consumption in beverage
  Arms: 1
Dietary Supplement: Novel dietary fiber — Oral consumption in beverage
  Arms: 2
Other: Placebo — Oral consumption in beverage
  Arms: Placebo beverage

SUMMARY:
This study will critically evaluate the effects of a novel dietary fiber administered to subjects at high risk for developing diabetes to determine if this intervention will improve insulin sensitivity compared to control product administration and, thus, decrease risk for developing diabetes.

The hypothesis is that consuming this novel fiber twice a day for 12 weeks will significantly decrease fasting plasma glucose, insulin and glycosylated hemoglobin values in pre-diabetic subjects (i.e. subjects with fasting plasma glucose levels 95-140 mg/dl at screening) compared to consumption of the control product.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of any racial/ethnic group; able to read, comprehend, and write English at a sufficient level to complete study-related materials
* Age: at least 30 and no more than 70 years at randomization into this trial
* BMI: 25-40 kg/m2 at randomization into this trial
* Fasting blood glucose: 95-140 mg/dl (for those with glucose 95-99mg/dl, must have history of gestational diabetes or first degree relative (parent or sibling) with history of diabetes; for those with glucose 100-125 mg/dl, will be enrolled as the primary target for recruitment; for those with glucose 126-140 mg/dl (asymptomatic diabetes), must not have prior diagnosis of diabetes and must not have prior treatment/pharmacotherapy for diabetes)
* Good general health as evidenced by the medical history
* Blood chemistry and urinalysis results within normal ranges or within an acceptable range determined by the physician on site and/or in consultation with the Medical Monitor
* Available and willing to participate in the study for up to 15 weeks
* Willing to follow a weight-maintaining Lifestyle diet throughout the 12 week trial, maintain physical activity patterns at baseline levels throughout the study period, and not add new exercise routines, dietary supplements, vitamins or other unusual food products
* Willing to consume two 16 oz beverages every day with meals for 12 weeks and able to transport the test article

Exclusion Criteria:

* Presence of any condition the Investigator believes would interfere with subject's ability to provide informed consent, comply with study instructions, or which might confound the interpretation of the study results or put the subject at undue risk
* Food allergy or sensitivity to any of the ingredients in the study product (e.g. Gluten sensitivity, celiac disease)
* Participation in another clinical trial that might interfere with this trial or exposure to any investigational agent within 30 days prior to first visit
* History of diabetes (subjects with a prior history of gestational diabetes may be enrolled if they had no pharmacologic treatment for diabetes since pregnancy)
* Treatment for diabetes or a related condition (e.g., polycystic ovary syndrome) with metformin, an oral agent, or insulin or other injections used for diabetes management
* Uncontrolled hypertension (i.e., systolic blood pressure >160 mm Hg, or a diastolic blood pressure >95 mmHg based on an average of 3 readings sitting)
* Fasting serum triglyceride value >250 mg/dl (since changes in triglyceride values can affect glucose homeostasis)
* Untreated hypothyroidism with a TSH > 1.5 times the upper limit of normal for the test laboratory with repeat value that also exceeds this limit
* Recent history of weight loss (>4 kg in the past 3 months) or a significant variation in weight (>4 kg in the past 3 months, for example, due to a medical condition such as pregnancy, or hormonal therapy)
* Use of medications or herbal remedies for weight loss (e.g., sibutramine, orlistat, amphetamines, phentermine, and ma huang) or use of these substances within the past 3 months
* Current or recent history (past 12 months) of drug, alcohol or chemical abuse. Alcohol abuse will be defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1.5 oz hard liquor)
* Pregnant, breast-feeding or female of child-bearing potential who is unwilling to commit to the use of a medically approved form of contraception throughout the study period.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Mean changes in fasting and post-glucose administration values for plasma glucose from baseline to end of study | 0, 6, 9, 12 weeks
Mean changes in fasting and post-glucose administration values for plasma insulin from baseline to end of study | 0, 6, 9, 12 weeks
Mean changes in blood HbA1c values from baseline to end of study | 0, 12 weeks

SECONDARY OUTCOMES:
Mean changes from baseline to end of study in HOMA | 0, 6, 9, 12 weeks
Percentage change and absolute change from baseline in body weight | 0, 3, 6, 9, 12 weeks
Mean changes from baseline in waist circumference | 0, 12 weeks
Mean changes in total body fat, lean tissue and abdominal fat as determined by DEXA [distribution or absolute changes] | 0, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Harold E Bays, MD, FACP, Principal Investigator — Louisville Metabolic and Atherosclerosis Research Center; Dale R Wilson, MD, CCFP(EM), FCFP, Principal Investigator — KGK Science Inc.
Locations (2):
- Louisville Metabolic and Atherosclerosis Research Center, Louisvile, Kentucky, United States
- KGK Synergize Inc., London, Ontario, Canada

REFERENCES:
- [Background] Weickert MO, Mohlig M, Schofl C, Arafat AM, Otto B, Viehoff H, Koebnick C, Kohl A, Spranger J, Pfeiffer AF. Cereal fiber improves whole-body insulin sensitivity in overweight and obese women. Diabetes Care. 2006 Apr;29(4):775-80. doi: 10.2337/diacare.29.04.06.dc05-2374. PMID 16567814
- [Background] Lu ZX, Walker KZ, Muir JG, Mascara T, O'Dea K. Arabinoxylan fiber, a byproduct of wheat flour processing, reduces the postprandial glucose response in normoglycemic subjects. Am J Clin Nutr. 2000 May;71(5):1123-8. doi: 10.1093/ajcn/71.5.1123. PMID 10799374
- [Background] Anderson JW, Kendall CW, Jenkins DJ. Importance of weight management in type 2 diabetes: review with meta-analysis of clinical studies. J Am Coll Nutr. 2003 Oct;22(5):331-9. doi: 10.1080/07315724.2003.10719316. PMID 14559925
- [Background] Behall KM, Scholfield DJ, Hallfrisch J. Comparison of hormone and glucose responses of overweight women to barley and oats. J Am Coll Nutr. 2005 Jun;24(3):182-8. doi: 10.1080/07315724.2005.10719464. PMID 15930484
- [Background] Jenkins AL, Jenkins DJ, Zdravkovic U, Wursch P, Vuksan V. Depression of the glycemic index by high levels of beta-glucan fiber in two functional foods tested in type 2 diabetes. Eur J Clin Nutr. 2002 Jul;56(7):622-8. doi: 10.1038/sj.ejcn.1601367. PMID 12080401
- [Background] Keenan JM, Goulson M, Shamliyan T, Knutson N, Kolberg L, Curry L. The effects of concentrated barley beta-glucan on blood lipids in a population of hypercholesterolaemic men and women. Br J Nutr. 2007 Jun;97(6):1162-8. doi: 10.1017/S0007114507682968. Epub 2007 Apr 20. PMID 17445284
- [Derived] Bays H, Frestedt JL, Bell M, Williams C, Kolberg L, Schmelzer W, Anderson JW. Reduced viscosity Barley beta-Glucan versus placebo: a randomized controlled trial of the effects on insulin sensitivity for individuals at risk for diabetes mellitus. Nutr Metab (Lond). 2011 Aug 16;8:58. doi: 10.1186/1743-7075-8-58. PMID 21846371